CLINICAL TRIAL: NCT03715270
Title: Prospective Non-randomized, Non-blinded, Convenience Sample to Evaluate the Surgical Imaging System
Brief Title: Evaluation of Tissue Oxygen Levels During Breast Reconstruction With a New Surgical Device
Acronym: Presygen™
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision to end study.
Sponsor: Christie Medical Holdings, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: #E-18-741
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Perfusion; Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- breast reconstruction surgery patients: Patients will be imaged with imaging device (Presygen™/si-1) during surgical procedure. Image surgical area. Surgical procedure will follow standard of care. No clinical decisions will be made on device readings. A surgeon will complete a survey regarding his assessment of the imaging device.
  Interventions: Device: Image surgical area

INTERVENTIONS:
Device: Image surgical area — Image surgical area
  Other Names: Questionnaire on ease of use and general opinion

SUMMARY:
This study is designed to evaluate the information provided to the clinicians by the surgical imaging device. It is also to gain insight on the user interface and how "user friendly" it is to the clinician.

DETAILED DESCRIPTION:
Over the last decade, objective ways of measuring tissue oxygen have been introduced into the medical arena and are being used more and more for assessing ischemic events in tissue. Handheld Doppler ultrasound, infrared thermography, polarized spectral imaging, laser Doppler perfusion imaging, and fluorescence imaging have all been used with some degree of success. However, only a few have gained universal acceptance. [1] Multispectral imaging (MSI) which uses near-infrared (NIR) light to measure tissue oxygen levels in superficial tissue is another method that has been successfully used to assess tissue flap health.

The objective of this study is to conduct an evaluation of superficial tissue with Presygen™/si-1 in various patient types for surgical imaging during breast reconstruction. In addition, participating surgeons will complete a structured survey regarding their assessment of Presygen™/si-1 work station during the surgical procedure.

Primary Goal: Evaluation of superficial tissue in various patient types for surgical imaging during breast reconstruction.

Secondary Goal: Surgeon assessment of surgical work station during surgery through a prepared questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for surgical intervention with breast reconstruction as part of the surgical plan
* 22 years of age or older;
* Able to understand and provide informed consent with HIPAA authorization.
* Able to read and understand in English.

Exclusion Criteria:

* Subjects who might need a legally-authorized representative
* Subjects who possess diminished mental capabilities
* Conditions that preclude imaging (excessive scarring, tattoos in surgical field, Fitzpatrick Scale VI)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing breast reconstruction surgery and meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Photographic, electronic and descriptive comparative analysis of superficial tissue oxygen saturation using Presygen™/si-1 for breast reconstruction subjects. | 24 hours.
  Quantitative measures of tissue oxygen saturation for discrete locations on superficial tissue.

SECONDARY OUTCOMES:
Quantitative survey providing surgeon assessment of work station during procedure. | 24 hours
  completion of basic questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Hospital and Medical Cetner, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pestana IA, Coan B, Erdmann D, Marcus J, Levin LS, Zenn MR. Early experience with fluorescent angiography in free-tissue transfer reconstruction. Plast Reconstr Surg. 2009 Apr;123(4):1239-1244. doi: 10.1097/PRS.0b013e31819e67c1. PMID 19337092
- [Result] Colwell AS, Craft RO. Near-infrared spectroscopy in autologous breast reconstruction. Clin Plast Surg. 2011 Apr;38(2):301-7. doi: 10.1016/j.cps.2011.03.014. PMID 21620154